CLINICAL TRIAL: NCT03710005
Title: Randomized Control Study Comparing Efficacy of a Dehydrated Cell and Protein Concentrate (dCPC) ("Ascent") Versus Corticosteroid
Brief Title: Efficacy of Dehydrated Cell and Protein Concentrate Versus Corticosteroid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA upregulation of dCPC.
Sponsor: StimLabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLAC-ORTHO-001
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascent Intervention Treatment (Experimental): Interventional treatment arm will receive Ascent dehydrated cell and protein concentrate injection
  Interventions: Procedure: Ascent
- Standard Treatment (Active Comparator): Standard treatment arm will receive a standard Corticosteroid injection
  Interventions: Procedure: Standard

INTERVENTIONS:
Procedure: Ascent — Dehydrated Cell and Protein Concentrate injection
  Arms: Ascent Intervention Treatment
Procedure: Standard — Standard corticosteroid injection
  Arms: Standard Treatment

SUMMARY:
To compare the efficacy of Ascent injection versus corticosteroid injection in treating knee osteoarthritis.

DETAILED DESCRIPTION:
To compare the functional outcomes in patients undergoing treatment of knee osteoarthritis using cortisone steroid injections (CSI) or a dehydrated cell and protein concentrate (dCPC) product, Ascent

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 20 years but less than 75 years old
* Both male and female (non-pregnant)
* Valid knee radiograph within 3 months of beginning treatment;
* Diagnosis of OA of the knee
* OA pain in the knee despite conservative measures
* Average daily VAS >= 3
* Off any NSAIDs for 1 week prior to injection, may then continue for no more than 5 consecutive days after injection
* Kellgren-Lawrence system of Grade II, III, or IV

Exclusion Criteria:

* Kellgren-Lawrence Grade I
* Tense effusion of the knee
* Significant valgus/varus deformities
* Viscosupplementation within 6 months
* Surgery in the knee within the past 6 months Systemic or intraarticular injection of costicosteroids in any joint within 3 months before screening
* Chronic opioid usage
* History of Leukemia or Lymphoma
* History of any autoimmune disorders and disease
* Immunosuppressive medications
* Active, suspected, or prior infection to the joint
* Vulnerable populations (pregnant women and breast-feeding women, cognitively impaired, prisoners, etc...)
* NSAIDs used within 1 week of the procedure
* History of bleeding disorders or inflammatory joint disease
* Patients who plan on becoming pregnant during study period

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Measuring changes in quality of life due to treatment, as assessed by patient reported survey. | 12 months
  The Quality of Life Survey is a patient-reported outcome measure divided into two parts. The first part of the Quality of Life questionnaire/survey will include 4 questions in which patients will be asked to evaluate their individual levels of knee problems (knee difficulty, knee confidence, and lifestyle modifications). Answers will be reported on a 5 point likert scale, in which higher scores indicate more severity, and lower scores indicate less severity. The second part of the questionnaire will include 6 categories (discomfort, mobility, self-care, anxiety, performance of activities, and sleeping). There will be 3 statements per category in which the patient is asked to indicate which statement best describes their current health. The questionnaire is scored by adding up the scores of each item to compute a total score.

SECONDARY OUTCOMES:
Measured change in pain: VAS | 12 months
  The Visual Analog scale is a patient-reported outcome measure. It will be presented numerically as an 11 point scale that will ask the patient to rate the severity of their pain on a scale form 0 to 10, which 10 being the most pain imaginable and 0 being the least (no pain). The numerical value will be reported based on the patient's response. The mean pain scores of each intervention group will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Oluseun Olufade, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Sports Medicine Complex, Brookhaven, Georgia
  - Emory At Dunwoody, Dunwoody, Georgia
  - Emory Orthopaedics and Spine Center, Johns Creek, Georgia
  - Emory at Smyrna, Smyrna, Georgia

REFERENCES:
- [Derived] Olufade O, Negron G, Berrigan W, Sirutis B, Whitley J, Easley K, Chen Y, Mautner K. Amniotic dehydrated cell and protein concentrate versus corticosteroid in knee osteoarthritis: preliminary findings. Regen Med. 2022 Jul;17(7):431-443. doi: 10.2217/rme-2022-0005. Epub 2022 May 19. PMID 35586982